CLINICAL TRIAL: NCT05687565
Title: Efficacy of Lauric Acid, a Dietary Fatty Acid, in Modifying the Latent Reservoir of HIV
Acronym: FATHIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)12/2022
Record Dates: First submitted 2022-12-13; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
Keywords: lauric acid; HIV; antiretroviral treatment
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Dietary supplementation
  Interventions: Dietary Supplement: Control group placebo
- Experimental group 1 (Experimental): 1.5 grams once daily during 48 weeks
  Interventions: Dietary Supplement: Experimental group 1 lauric acid
- Experimental group 2 (Experimental): 3 grams once daily during 48 weeks
  Interventions: Dietary Supplement: Experimental group 2 lauric acid

INTERVENTIONS:
Dietary Supplement: Control group placebo — Dietary suplementation
  Arms: Control group
Dietary Supplement: Experimental group 1 lauric acid — Lauric acid 1.5 grams once daily
  Arms: Experimental group 1
Dietary Supplement: Experimental group 2 lauric acid — Lauric acid 3 grams once daily
  Arms: Experimental group 2

SUMMARY:
Dietary lauric acid supplementation could have a significant impact on the HIV reservoir in antiretroviral-treated patients by inducing HIV viral transcription in latently infected cells and preserving the HIV-specific immune response, without causing toxicity.

Design: Pilot, randomized, placebo-controlled, patient-blind study. Patients ≥18 years old with HIV-1 receiving stable ART (no change in ART for at least 6 months) and a serum HIV RNA load of < 50 RNA copies/mL for at least 2 years and with a CD4 T cell count >300 cells/μl will be randomized 1:1:1 to dietary supplementation with placebo (controlled group) or lauric acid 1.5 g once daily (experimental group 1) or with lauric acid 3 g once daily (experimental group 2) for 24 consecutive weeks.

Primary objective: To assess the effect of dietary lauric acid supplementation, compared with placebo, on the reactivation of HIV transcription in latently infected CD4 T cells in HIV-infected patients on suppressive antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected men or women ≥18 years old
* Not having interrupted current antiretroviral treatment at least 6 months before the screening visit.
* Acceptable stable ART regimens prior to screening include 2 more NRTIs: INI or NNRTI or boosted PI.
* Documented prior evidence of at least 2 years prior to enrollment with a serum HIV RNA load of <50 RNA copies/ml (viral load of >50 copies but <200 is allowed).
* Plasma HIV-1 RNA <50 c/ml at screening visit.
* CD4 T cell count > 300 cells/µL at screening visit.

A woman may be eligible to enroll and participate in the study if:

* Not pregnant, not of childbearing potential or physically unable to become pregnant
* You are of childbearing potential with a negative pregnancy test at the screening visit and agree to use contraception to prevent pregnancy.

Exclusion Criteria:

* Have suffered any significant acute illness in the last 8 weeks.
* Having been diagnosed in the past or present with an AIDS-defining illness
* Previous CD4 T cell count <200 cells/μL.
* Having suffered an infection with Hepatitis B or C
* Having any disease or condition that in the investigator's opinion is not appropriate for the patient's participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Effective of lauric acid in HIV | 48 weeks
  Number of patients on a lauric acid diet presenting a response on the reactivation of HIV transcription in CD4 T cells.

SECONDARY OUTCOMES:
Effective of lauric acid on the size of the latent HIV-1 reservoir in CD4 T cells | 48 weeks
  To dertermine the effetive of lauric acid on the size of the latent HIV-1 reservoir in CD4 T cells
Effective of lauric acid on the production of HIV-1 viral | 48 weeks
  To dertermine the effetive of lauric acid on on the production of HIV-1 viral (viral load)
Effective of lauric acid on the size of the HIV-1 reservoir in intestinal tissue | 48 weeks
  To dertermine the effetive of lauric acid on the size of the HIV-1 reservoir in intestinal tissue
Evaluate Lauric acid plasmatic levels | 48 weeks
  To evaluate Lauric acid with high performance liquid chromatography (HPLC).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Vall d´Hebron, Barcelona, Spain